CLINICAL TRIAL: NCT06948617
Title: Digital and Conventional Impression Techniques: What Influences Children's Preferences?
Brief Title: Children's Preferences on Digital and Conventional Impression Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 333-333-11
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Dental Impressions
Keywords: dental impression; digital intraoral scanner; alginate; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children aged between 5-11 who need space maintainer or orthodontic treatments (Experimental)
  Interventions: Device: digital intraoral scanner; Device: Alginate Impression

INTERVENTIONS:
Device: digital intraoral scanner — Alginate impressions were obtained with an irreversible hydrocolloid impression material (Cavex Impressional; Cavex Holland, Haarlem, The Netherlands) and standard plastic trays. For each impression, the time required to mix the material and complete a full-mouth (maxillary and mandibular arches) impression was recorded.
Device: Alginate Impression — Alginate impressions were obtained with an irreversible hydrocolloid impression material (Cavex Impressional; Cavex Holland, Haarlem, The Netherlands) and standard plastic trays. For each impression, the time required to mix the material and complete a full-mouth (maxillary and mandibular arches) impression was recorded.

SUMMARY:
The goal of this crossover study is to compare children's perceptions and preferences regarding digital and conventional impression techniques in the 5- to 11-year-old age group. The main questions it aims to answer are

* Which impression methods do kids prefer?
* What influences kids' perception of impression methods?

Dental impressions will be obtained using both the conventional alginate impression (CAI) (Cavex ColorChange; Cavex Holland BV, Haarlem, the Netherlands) and digital intraoral scanning procedure (DIS) (3Shape TRIOS Color, 3Shape, Copenhagen, Denmark). After each procedure, patients will score their perceptions using a Modified Impression Perception Test, a 5-point Likert scale, for gag reflex, queasiness, difficulty breathing, uncomfortable feeling, pain perception, chairside time, and stress levels. Dental anxiety will be assessed using the Visual Anxiety Scale (1-10). Children will also be asked about their preferences and reasons in one or two sentences. Content analysis will be performed on answers to open-ended questions. Statistical analysis will be done using Fisher's Exact test.

ELIGIBILITY:
Inclusion Criteria:

* No prior exposure to either digital or conventional impression techniques
* Absence of temporomandibular joint disorders and periodontal disease
* Cleft lip and/or palate, or other significant craniofacial anomalies
* No current use of psychiatric or neuropathic medications

Exclusion Criteria:

* Individuals with a known history of dental anxiety or a pronounced gag reflex

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Modified Children Perception test | one year
  After the each impression proscedure, to evaluate children's perspectives on the impression techniques, the perception questionnaire used in Burhardt's study was adapted for this research.5 The questionnaire was translated into Turkish to ensure cultural and linguistic appropriateness. The translated version underwent content validation through expert review to ensure its relevance and appropriateness for the target population. The perception questionnaire used in this study aimed to measure gag reflex, queasiness, difficulty to breathe, discomfort, time perception, stress, pain. Accordingly, 8 questions with 5-point Likert scale responses ranging from "strongly agree" to "strongly disagree" were included (Figure-1). Additionally, the Visual Anxiety Scale (VAS) was employed to measure overall discomfort. For the VAS results, children were asked to score their perceived discomfort on a scale from 0 (no discomfort) to 10 (extreme discomfort).

SECONDARY OUTCOMES:
Responses to open-ended questions | one year
  After completing both of the impression proscedure, children were asked two questions regarding their preference: one closed-ended question "Which method did you prefer?" and one open-ended follow-up question "Why did you prefer this method?". The latter was used for thematic content analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University School of Dentistry, Department of Pediatric Dentistry, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data includes personel data of the participants.

REFERENCES:
- [Background] Yilmaz H, Aydin MN. Digital versus conventional impression method in children: Comfort, preference and time. Int J Paediatr Dent. 2019 Nov;29(6):728-735. doi: 10.1111/ipd.12566. Epub 2019 Aug 13. PMID 31348834